CLINICAL TRIAL: NCT02252094
Title: Ultra-protective Pulmonary Ventilation Supported by Low Flow Extracorporeal Carbon Dioxide Removal (ECCO2R) and Prone Positioning for ARDS; a Pilot Study.
Brief Title: Ultra-protective Pulmonary Ventilation Supported by Low Flow ECCO2R for Severe ARDS
Acronym: U-Protect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device no longer available in Singapore
Sponsor: National University Health System, Singapore (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Matthew COVE, Matthew COVE, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRC/TA/0015/2013
Record Dates: First submitted 2014-09-17; First posted 2014-09-29 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional lung protective ventilation (Active Comparator): Lung protective ventilation (6ml/kg predicted body weight). All other interventions per intensive care unit standardised ARDS management protocol
  Interventions: Other: Conventional Lung Protective Ventilation
- Ultra-protective ventilation (Experimental): Ultra-protective ventilation (</= 3ml/kg predicted body weight) targeting plateau pressure of </= 25 cmH2O, supported by Prismalung. All other intervention per intensive care unit standardised ARDS management protocol
  Interventions: Device: Prismalung; Other: Ultra-protective ventilation

INTERVENTIONS:
Device: Prismalung — Prism lung (Baxter Healthcare/Gambro Lund, Sweden) is an extracorporeal carbon dioxide removal device. It removes blood through a double lumen catheter and pumps it through a hollow fiber gas exchange cartridge which is impervious to fluid. Carbon dioxide diffuses out, down a concentration gradient which is maintained by sweep gas flowing through the centre of the hollow fibres. The decarboxylated blood is returned to the patient through the double lumen catheter.
  Other Names: Low flow extracorporeal carbon dioxide removal; Respiratory Dialysis
  Arms: Ultra-protective ventilation
Other: Ultra-protective ventilation — Ventilation with </= 3ml/kg predicted body weight
  Arms: Ultra-protective ventilation
Other: Conventional Lung Protective Ventilation — Ventilation with 6ml/kg predicted body weight
  Arms: Conventional lung protective ventilation

SUMMARY:
This study evaluates the use of ultra-protective ventilation, where very low ventilation volumes are used, in patients with severe acute respiratory distress syndrome (ARDS) meeting criteria to nurse in the prone position. Half the patients will receive ultra-protective ventilation support by extracorporeal carbon dioxide removal, while the other half will receive conventional lung protective ventilation.

DETAILED DESCRIPTION:
Current best practices for management of severe ARDS include lung protective ventilation and nursing in the prone position. However, the best lung protective strategy is not currently established and using smaller ventilation volumes than standard lung protective ventilation suggest lung recovery is improved.

Application of smaller ventilation volumes requires extracorporeal carbon dioxide removal, using a device similar to a dialysis to remove carbon dioxide directly from the blood. One such device in the Prismalung, it removes blood through a catheter, much like a dialysis catheter, pumps it through a gas exchange cartridge which removes carbon dioxide. The gas exchange cartridge functions in a similar way to a dialysis filter, except it allow gases to pass through, unlike dialysis filters which allow passage of fluid and small molecules.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to MICU with respiratory failure and intubated
* ARDS criteria per Berlin definition
* PaO2:FiO2 ratio ≤ 200 mmHg for > 6 hours with FiO2 ≥0.5
* Expected to require mechanical ventilation for >48 hours
* Reversible disease

Exclusion Criteria:

* Anticoagulation contraindicated
* Proven HIT
* Unable to obtain central venous access
* Refractory hypoxia (PaO2:FiO2 ≤80 after recruitment and proning) or other indication for ECMO
* Home oxygen use
* Severe COPD
* Interstitial lung disease
* > 7 days of mechanical ventilation
* Immunocompromised patient (bone marrow, untreated HIV, PJP)
* Advanced malignancy with life expectancy ≤ 6months

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Plateau Pressure | Duration of ventilation for severe ARDS, expected average time 10 days
  Ability to achieve a plateau pressure of </=25 cmH20 in the intervention arm

SECONDARY OUTCOMES:
Length of stay in ICU stay | Duration of patient stay in ICU, expected average stay 2 weeks
Length of hospital stay | Duration of patient stay in hospital
Mortality | Monitored for 3 months
  ICU mortality, hospital mortality, 30 day, 60 day and 90 day mortality
Cardiac Imaging | One data set per patient during first 72 hours
  Echocardiogram data will be collected before prone position, after prone positioning and following initiation of ultra-protective ventilation
Extracorporeal carbon dioxide removal related complications | Duration of severe ARDS, expected average time frame 10 days
  Complications or adverse events related to ECCO2R and associated anticoagulation
Ventilator free days | 28 days
All severe adverse events | Duration of ICU stay (anticipate average stay 1-2 weeks)
Number of patient meeting proning criteria in each group | Duration of ICU stay
Ability to successfully prone | Duration of ICU stay
Incidence of dialysis in ICU, and ability to successfully initiate | Duration of ICU stay
Incidence of referrals for ECMO | Duration of ICU stay
Rate and reasons for declining consent to study participation | First 48 hours
Enrolment rates | First 48 hours
Lung recruitability | Duration of ICU stay
Ventilation parameters | Duration of mechanical ventilation
  Data download from mechanical ventilation
Ventilator associated pneumonia rates | Duration of ICU stay
Barotrauma complications | Duration of ICU stay
Biomarkers of Pulmonary Inflammation | Day 0, 4 and 7
  Serum will be drawn and stored for pulmonary biomarkers analysis at the above time points

CONTACTS AND LOCATIONS:
Overall Officials: Matthew E Cove, MBChB, Principal Investigator — National University Health System
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terragni PP, Del Sorbo L, Mascia L, Urbino R, Martin EL, Birocco A, Faggiano C, Quintel M, Gattinoni L, Ranieri VM. Tidal volume lower than 6 ml/kg enhances lung protection: role of extracorporeal carbon dioxide removal. Anesthesiology. 2009 Oct;111(4):826-35. doi: 10.1097/ALN.0b013e3181b764d2. PMID 19741487
- [Background] Bein T, Weber-Carstens S, Goldmann A, Muller T, Staudinger T, Brederlau J, Muellenbach R, Dembinski R, Graf BM, Wewalka M, Philipp A, Wernecke KD, Lubnow M, Slutsky AS. Lower tidal volume strategy ( approximately 3 ml/kg) combined with extracorporeal CO2 removal versus 'conventional' protective ventilation (6 ml/kg) in severe ARDS: the prospective randomized Xtravent-study. Intensive Care Med. 2013 May;39(5):847-56. doi: 10.1007/s00134-012-2787-6. Epub 2013 Jan 10. PMID 23306584